CLINICAL TRIAL: NCT01829893
Title: Open Label, Randomized Comparative Study to Evaluate the Pharmacokinetic Characteristics Between Coadministered Finasteride Tablet and Tamsulosin HCl Tablet and GL2701 Capsule, in Healthy Subjects
Brief Title: PK Comparison of GL2701 With Finasteride and Tamsulosin in Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: GL Pharm Tech Corporation (Industry)
Responsible Party: Principal Investigator, Ji-Young Park, Associate Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: GP-FITAM-104
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2011-12

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: Benign Prostatic Hyperplasia (BPH); pharmacokinetics; bioequivalence; finasteirde; tamsulosin
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Finasteride; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference arm (Active Comparator): Treated with Reference (in combination of 0.2mg tamsulosin and 5mg finasteride) Intervetion: In combination of 0.2mg finasteride and 5mg tamsulosin simultaneously
  Interventions: Drug: In combination of 0.2mg finasteride and 5mg tamsulosin
- Test arm (Experimental): Treated with Test formulation (single pill combination of 0.2mg finasteride and 5mg tamsulosin) Intervention : GL2701 capsule
  Interventions: Drug: GL2701 capsule

INTERVENTIONS:
Drug: In combination of 0.2mg finasteride and 5mg tamsulosin — oral medication with 240 mL water
  Other Names: GL2701 capsule
  Arms: Reference arm
Drug: GL2701 capsule — oral medication with 240 mL water
  Other Names: Harunal-D (tamsulosin 0.2mg); Prosca (Finasteride 5 mg)
  Arms: Test arm

SUMMARY:
To compare the relative bioavailability and pharmacokinetic characteristics of a newly single pill combination of finasteride and tamsulosin with a conventional combination of finasteride and tamsulosin in healthy subjects with a single dose, randomized, open-label, 2-sequence -2period crossover study.

DETAILED DESCRIPTION:
This single dose, open label, balanced, randomized, two-treatment, two-period, two-sequence, crossover study was conducted to compare the relative bioavailability and pharmacokinetic characteristics of a newly developed formulation with a conventional formulation in healthy subjects.

For this, a single-center, randomized, single-dose, open-label, 2-period and 2-sequence crossover study with a 14-day washout period was conducted in 26 healthy volunteers. Plasma samples for the analysis of finasteride/tamsulosin were collected up to 48 h after drug administration. Participants received either reference (in combination of of 0.2mg tamsulosin and 5mg finasteride) or test drug formulation (single pill combination of 0.2mg tamsulosin and 5mg finasteride) in the first period and the alternative formulation in the second period. Plasma concentrations of both tamsulosin and finasteride were determined by validated high-performance liquid chromatography coupled to tandem mass spectrometry detection. Pharmacokinetic parameters, including Cmax and AUC, were determined by noncompartmental analysis. Analysis of variance (ANOVA) was carried out using log-transformed Cmax and AUC, and the mean ratios and their 90% confidence intervals (CI) were calculated. According to regulatory requirements set forth by Korea and the US Food and Drug Administration, products meet the criteria for bioequivalence if the 90% CIs of the mean ratios for Cmax and AUC are within the range of 0.80 to 1.25.

ELIGIBILITY:
Inclusion Criteria:

* Males age 20 to 45 years
* Body weight > 50 kg with 18~29 kg/m2 body mass index (BMI)
* Signed and dated informed consent form which meets all criteria of current FDA and KFDA regulations

Exclusion Criteria:

* subjects with acute conditions.
* presence of history affecting ADME
* Clinically significant history or current evidence of a hepatic, renal, gastrointestinal, or hematologic abnormality
* Hepatitis B, hepatitis C, or HIV infection revealed on the laboratory findings
* Any other acute or chronic disease
* A history of hypersensitivity to donepezil
* A history of alcohol or drug abuse
* Participation in another clinical trial within 3 months
* smoked >10 cigarettes daily
* consumption over 5 glasses daily of beverages containing xanthine derivatives
* use of any medication having the potential to affect the study results within 10 days before the start of the study.
* AST or ALT > 1.25 of upper normal limit
* total bilirubin > 1.5 of upper normal limit
* systolic blood pressure < 90 mmHg
* calculated CLcr using Cockroft-Gault equation < 50 mL/min

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Finasteride and Tamsulosin pharmacokinetics (Cmax and AUC) | 48 hr

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Young Park, MD, PhD, Principal Investigator — Department of Clinical Pharmacology & Toxicology, Anam Hospital, Korea University College of Medicine
Locations (1):
- Clinical trial center of Anam Hospital, Seoul, South Korea